CLINICAL TRIAL: NCT01687608
Title: A Phase 1/2 Open-Label, Single Ascending Dose Trial of a Self-Complementing Optimized Adeno-associated Virus Serotype 8 Factor IX Gene Therapy (AskBio009) in Adults With Hemophilia B
Brief Title: Open-Label Single Ascending Dose of Adeno-associated Virus Serotype 8 Factor IX Gene Therapy in Adults With Hemophilia B
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Baxalta now part of Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AskBio009-101; 231401 (Other: Sponsor)
Record Dates: First submitted 2012-08-27; First posted 2012-09-19 (Estimated); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Hemophilia B
Keywords: Hemophilia B; factor IX deficiency; gene therapy
MeSH Terms: conditions — Hemophilia B | interventions — BAX 335

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AskBio009 Dose Escalation (Experimental): Single Dose of a Self-Complementing Optimized Adeno-associated Virus (AAV) Serotype 8 Factor IX Gene Therapy
  Interventions: Biological: AskBio009

INTERVENTIONS:
Biological: AskBio009 — Single dose IV injection
  Other Names: BAX 335

SUMMARY:
The purpose of this study is to evaluate the safety of single ascending IV doses of a Factor IX (FIX) Gene Therapy in up to 16 Adults with Hemophilia B.

DETAILED DESCRIPTION:
Hemophilia B is a genetic X-linked bleeding disorder caused by a deficiency in blood-clotting Factor IX (FIX) activity. FIX is synthesized in the liver and circulates in the blood as a proenzyme. Current treatment for hemophilia B is based on replacement of the deficient FIX with IV injections of recombinant FIX protein prophylactically or as needed to treat bleeding episodes. This clinical program will test a gene transfer approach involving the use of a gene delivery vector carrying a FIX gene. This first-in-humans study is intended to evaluate the safety, kinetics, and if possible, the dose of AskBio009 required to achieve stable plasma FIX activity between 10% and 40% of normal activity.

ELIGIBILITY:
Inclusion Criteria:

* Males age 18-75 years, inclusive
* Established hemophilia B with ≥3 hemorrhages per year requiring treatment with exogenous FIX OR use of FIX prophylaxis because of history of frequent bleeding episodes
* Plasma FIX activity ≤2% (<1% for first cohort; then per protocol)
* Negative for active Hepatitis C virus (HCV), defined as Hepatitis C virus antibody negative and negative (undetectable) PCR test for plasma Hepatitis C virus ribonucleic acid (RNA) OR if Hepatitis C virus antibody positive must have ≥2 consecutive negative (undetectable) PCR tests for plasma HCV RNA at least 3 months apart, and negative at screening

Exclusion Criteria:

* Family history of inhibitor to FIX protein or personal laboratory evidence of having developed inhibitors to FIX protein at any time (>0.6 Bethesda Units on any single test)
* Documented prior allergic reaction to any FIX product
* Detectable AAV8 neutralizing antibodies
* Markers of hepatic inflammation or overt or occult cirrhosis as evidenced by one or more of the following:

  * Platelet count <175,000/μL
  * Albumin ≤3.5 g/dL
  * Total bilirubin >1.5 x ULN and direct bilirubin ≥0.5 mg/dL
  * Alkaline phosphatase >2.0 x ULN
  * ALT or AST >2.0 x ULN (except for subjects who are HIV infected)
  * Liver biopsy in the past indicating moderate or severe fibrosis (Metavir staging of 2 or greater)
  * History of ascites, varices, variceal hemorrhage or hepatic encephalopathy

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-02-11 (Actual); Primary Completion 2030-01-17 (Estimated); Study Completion 2030-01-17 (Estimated)

PRIMARY OUTCOMES:
Number of patients experiencing treatment-related adverse events by dose group | Infusion to Week 3 and Infusion to end of study
Change from baseline in clinical laboratory evaluations | Change from baseline at week 3 and change from baseline at the end of study

SECONDARY OUTCOMES:
Changes from Baseline in FIX activity levels, FIX protein levels, and Bleeding Episode Severity & Frequency | At multiple timepoints from pre-dose through up to 5 years post-dose
Immune Response to AskBio009 | At multiple timepoints from pre-dose through up to 5 years post-dose
Detection of AskBio009 genomes in blood, saliva, urine, stool, and semen | At multiple timepoints from pre-dose through up to 1 years post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Shire
Locations (15):
- United States (15):
  - Orthopaedic Hemophilia Treatment Center, Los Angeles, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - University of California Davis Medical Center, Sacramento, California
  - University of California at San Diego Medical Center, San Diego, California
  - U of Colorado School of Medicine, Hemophilia & Thrombosis Treatment Center, Aurora, Colorado
  - Emory University, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Children's Hospital of Boston, Boston, Massachusetts
  - University of Minnesota, Masonic Clinical Research Unit, Clinical and Translational Science Institute, Minneapolis, Minnesota
  - Mount Sinai Medical Center, New York, New York
  - The Hemophilia Center, Oregon Health and Science University, Portland, Oregon
  - Medical University of South Carolina, Charleston, South Carolina
  - Gulf States Hemophilia and Thrombosis Center, Houston, Texas
  - Bloodworks Northwest, Seattle, Washington
  - BloodCenter of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Konkle BA, Walsh CE, Escobar MA, Josephson NC, Young G, von Drygalski A, McPhee SWJ, Samulski RJ, Bilic I, de la Rosa M, Reipert BM, Rottensteiner H, Scheiflinger F, Chapin JC, Ewenstein B, Monahan PE. BAX 335 hemophilia B gene therapy clinical trial results: potential impact of CpG sequences on gene expression. Blood. 2021 Feb 11;137(6):763-774. doi: 10.1182/blood.2019004625. PMID 33067633
- [Derived] Weber A, Engelmaier A, Voelkel D, Pachlinger R, Scheiflinger F, Monahan PE, Rottensteiner H. Development of Methods for the Selective Measurement of the Single Amino Acid Exchange Variant Coagulation Factor IX Padua. Mol Ther Methods Clin Dev. 2018 Jun 28;10:29-37. doi: 10.1016/j.omtm.2018.05.004. eCollection 2018 Sep 21. PMID 30003118
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/find-a-trial?idFilter=%5B%22AskBio009-101%22%5D